CLINICAL TRIAL: NCT05339841
Title: Digital Strategies in Primary Cardiovascular Prevention in the Italian Population
Brief Title: Italian Digital Primary Cardiovascular Prevention Study
Acronym: CV-PREVITAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Istituto Auxologico Italiano (Other); Humanitas Hospital, Italy (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); IRCCS Multimedica (Other); Neuromed IRCCS (Other); IRCCS Policlinico S. Donato (Other); Istituti Clinici Scientifici Maugeri SpA (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); Ospedale Policlinico San Martino (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); IRCCS San Raffaele Roma (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R1256/20-CCM 1319; RCR-2019-23669116_001 (Other Grant/Funding Number: MINISTERO DELLA SALUTE)
Record Dates: First submitted 2021-09-09; First posted 2022-04-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy Population
Keywords: CV primary prevention; CV risk factors; Hypertension; Diabetes; Hypercholesterolemia; Lifestyle behaviours; Digital Health; mHealth; Mobile app; Health empowerment; Primary care
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in two parallel groups:" intervention group" and "usual care". In the setting of general medicine, the procedure randomises the general practitioners (GPs) assuring that in each recruiting centre the number of GPs assigned to the control group (usual care) is balanced with that assigned to the intervention group. In the setting of community pharmacies, the procedure randomises the pharmacies assuring that in each geographic area the number of pharmacies assigned to the control group and is balanced with that assigned to the intervention group. In the setting of IRCCS the procedure directly randomises the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Subjects monitored following usual-care.
- Intervention group (Experimental): Subjects in the intervention group, in addition to usual-care, will download a mHealth App that contains educational information promoting healthy lifestyle behaviours. The participant will be also able to self-monitor his/her clinical status regarding hypertension, diabetes or hypercholesterolemia.
  Interventions: Other: Mobile health application

INTERVENTIONS:
Other: Mobile health application — The mHealth app delivers a personalized support program of digital health. Specifically, using ad hoc designed algorithms which uses the data self-reported by the subject and/or collected by the recruiter at baseline, the App delivers periodic messages with advice, motivational reminders and support to improve lifestyle habits and risk factor control.
  Other Names: mHealth app
  Arms: Intervention group

SUMMARY:
The CV-PREVITAL study is a randomised clinical trial (RCT) controlled versus usual-care designed to compare the effectiveness of a mobile health (mHealth) intervention with that of usual care in reducing specific cardiovascular (CV) risk factors (in the short term) and the occurrence of vascular events (in the long term). Promoted by the Italian Network of Cardiology (ICN, a cardiovascular research network promoted by the Italian Ministry of Health), in collaboration with the Consorzio Sanità (Co.S., an Italian consortium of general practitioners), CV-PREVITAL aims to develop an innovative model of cardiovascular primary prevention and to validate it in a very large sample of subjects and in 'real life' conditions.

DETAILED DESCRIPTION:
CV-PREVITAL is an RCT investigating whether an mHealth application (App) provided on top of usual care, can improve lifestyle habits and CV risk factor control in the short-term, and the incidence of major CV events in the long- term. Participants undergo two clinical visits, the first at baseline and the second after 12 months. During these visits, total cholesterol, HDL, LDL, triglyceride, HbA1c, blood pressure, heart rate, BMI and waist circumference are measured. In addition, using questionnaires provided digitally, participants self-report data on the following topics: adherence to the Mediterranean diet, salt intake, alcohol consumption, physical activity, current and previous smoking history, psychosocial profile, and sleep quality. Demographic information, including education, socio-economic status and ethnic origin are also obtained at baseline. Subjects in the intervention group also receive the credentials to download the App, which contains educational information on cardiovascular risk factors, diet, physical activity, lifestyle and psycho-behavioral aspects. Using ad hoc designed algorithms, the App delivers personalized prevention programs based on periodic messages providing advice, motivational reminders and support to improve lifestyle and risk factor control. When at baseline high levels of blood pressure, blood glucose or cholesterol are detected, the App support the participant in self-monitoring the clinical changes of such variables during the follow up. The efficacy of the intervention is evaluated at the12th month using a cardiovascular risk score developed ad hoc in an Italian population (Modified Moli-Sani Score). The ability of the intervention to maintain its effect over time and its effectiveness in improving clinical outcomes are assessed at the 7th year of follow-up. The cost-effectiveness of the intervention is also evaluated at the 7th year.

The study envisages the recruitment of 82,800 participants (aged ≥45y) nationwide. Of these, 50,000 are selected among those who daily access the GPs ambulatories associated to the Co.S. consortium. In order to assess whether the scheduled mHealth intervention can be effective also in settings different from the primary care, several specific cohorts in primary prevention are also enrolled by specialized units belonging to Scientific Institutes for Research, Hospitalization and Health Care (Italian acronym IRCCS). These cohorts include 32,800 subjects in total. Specifically, the UO-1 (IRCCS Cardiologico Monzino in Milan) enrolls 5,000 participants selected among citizens attending to community pharmacies; the UO-2 (IRCCS Auxologico in Milan) enrolls 5,000 subjects, 1,500 of which belonging to the Centre for Sleep Medicine; the UO-3 (IRCCS Humanitas in Milan) enrolls 2,000 subjects attending the institution; the UO-4 (IRCCS Mario Negri in Milan) does not recruit any subject but provides scientific and organizational support for the enrolment carried out by Co.S.; the UO-5 (IRCCS MultiMedica in Milan) enrolls 1,000 subjects with diabetes and 2,000 subjects from the general population; the UO-6 (IRCCS Neuromed in Pozzilli) enrols 10,000 subjects from the Neuromed clinical research centres; the UO-7 (IRCCS San Donato in Milan) enrolls 1,000 subjects selected among its own employees; the UO-8 (IRCCS Maugeri in Pavia) enrolls 1,000 subjects selected among its own employees; the UO-9 (IRCCS ISMETT, Mediterranean Institute for Transplantation and Advanced Specialized Therapies, in Palermo) enrolls 150 subjects who undergoes a physical activity program; the UO-10 (IRCCS San Martino in Genoa) enrolls 2,000 male subjects from the Municipality of Genoa; the UO-11 (IRCCS Ca' Granda of Milan) enrolls 2,000 blood donors afferent to its own Department of Transfusion Medicine and Hematology (DMTE); the UO-12 (IRCCS Gemelli in Rome) enrolls 1,000 subjects attending to the outpatient clinics of the Non-Invasive Cardiology Diagnostic Unit, of the Centre for Hypertension, and of the Centre for Endocrine and Metabolic Diseases; the UO-13 (IRCCS San Matteo in Pavia) enrolls 500 subjects selected among asymptomatic relatives of patients attending to the Policlinico San Matteo for cardiology reasons; the UO-14 (IRCCS San Raffaele in Rome) enrolls 150 subjects selected among its own employees.

Baseline data of the 82,800 participants and 1- and 7-years outcomes are also used to develop and validate a new algorithm for cardiovascular risk estimation. The new algorithm is developed by identifying among alcohol intake (as assessed by PREDIMED questionnaire), salt intake (as assessed by MiniSal questionnaire), perceived stress (as assessed by perceived stress scale (PSS), anxiety and depression (as assessed by Patient Health Questionnaire 4; PHQ 4), Locus of control (as assessed by Multidimensional Health Locus of Control scale, MHLCS), General Self Efficacy (as assessed by General Self Efficacy Scale; GSE), Risk propensity (as assessed by Risk Propensity Scale; RPS), and sleep quality (as assessed by Pittsburgh Sleep Quality Index) those variables that significantly improve the predictive power of the modified Moli-Sani algorithm.

The CV-PREVITAL trial also envisages a series of ancillary studies that are conducted by the various IRCCSs on the subjects already participating in the main study. Each ancillary study has its own protocol and aims, and foresees the evaluation of the role of further biomarkers relevant in the assessment of cardiovascular risk. The sub-study aims, outcomes information and time frame are described below. Baseline data of many ancillary studies are used to identify conventional and emerging determinants of specific cardiometabolic diseases. Specifically: a) the IRCCS Monzino analyses with multivariable approaches determinants and factors predisposing to diabetes status as assessed by Framingham diabetes score; b) the IRCCS Auxologico will apply additional elements for risk stratification including biomarkers high sensitive C-reactive protein (hs-CRP), Troponin I, N-terminal pro-brain natriuretic peptide (NT-proBNP), as well as 24 h ABPM (Ambulatory Blood Pressure Monitoring) derived variables; c) the IRCCS Humanitas analyses the frequency of genetic polymorphisms related to severe coronary calcification of its own cohort to identify genetic determinants of severe coronary calcification; d) the IRCCS MultiMedica analyses with multivariable approaches anthropometric (e.g. weight, height, BMI), biochemical data (e.g. lipid profile) and specific genetic disorders (e.g. presence of causative mutations in known genes involved in dyslipidemia) to identify determinants predisposing to dyslipidemia, hypertension and diabetes; e) the IRCCS Neuromed analyses with multivariable approaches determinants of dietary changes in the CV-PREVITAL Neuromed sub-study cohort; f) the Istituti Clinici Scientifici Maugeri IRCCS analyses baseline data of its own cohort with multivariable approaches to identify determinants of organ damage such as coronary silent ischemia, ankle brachial index, coronary calcium score and carotid ultrasound as well as Genetic and epigenetic (DNA and RNA) and other chemical determinants and factors predisposing to atherosclerotic diseases; g) the IRCCS Ca' Granda performs a 7 years validation of new monogenic and polygenic cardiovascular risk scores in its own primary prevention cohort. To this aim the study cohort is genotyped with GWAS and Whole Exome Sequencing (WES) for genetic factors influencing intracellular lipid handling (PNPLA3 I148M, TM6SF2 E167K, GCKR P446L, MBOAT7). Epigenetic variables indicated in the literature as early predictors of cardiovascular injury and cardiovascular events are also investigated. In addition to the characterization of genetic variants in known associated genes, the genomic characterization will allow the validation of candidate risk variants in genes reported to influence cardiovascular damage, the identification of potentially new candidate variants, and the calculation of polygenic cardiovascular risk scores and of their possible application to disease risk stratification in the Italian population; h) the IRCCS San Matteo develops new monogenic and polygenic scores and validates existing scores for the risk assessment of developing diabetes, hypertension and hypercholesterolemia.

Beyond the specific aims of the single sub-studies, a relevant goal common to all sub-studies is the collection of biological samples for the multisite biobank of the ICN.

The full list of approving body and approval number/ID of CV-PREVITAL studies is reported below.

Parent study: Approval Number: R1256/20-CCM 1319; Board Name: Comitato Etico degli IRCCS Istituto Europeo di Oncologia e Centro Cardiologico Monzino.

Ancillary studies of Monzino: Approval Number: R1579/21-CCM 1677 and R1617/22-CCM 1723; Board Name: Comitato Etico degli IRCCS Istituto Europeo di Oncologia e Centro Cardiologico Monzino.

Ancillary study of Istituto Auxologico Italiano: Approval Number: 2022_03_08_06; Board Name: Comitato Etico dell'IRCCS Istituto Auxologico Italiano.

Ancillary study of Humanitas: Approval Number: 2860; Board Name: Comitato Etico Indipendente dell'Istituto Clinico Humanitas.

Ancillary study of Multimedica: Approval Number: MM: 472.2021; Board Name: Comitato Etico IRCCS Multimedica - Sezione del Comitato Etico Centrale IRCCS Lombardia.

Ancillary study of Neuromed: Approval: Session of 28/09/2020; Board Name: Comitato Etico dell'Istituto Neurologico Mediterraneo Neuromed.

Ancillary study of San Donato: Approval Number: 197/INT/2021; Board Name: Comitato Etico IRCCS Ospedale San Raffaele.

Ancillary study of Maugeri: Approval Number: 2575 CE; Board Name: Comitato Etico degli Istituti Clinici Scientifici Maugeri.

Ancillary study of ISMETT: Approval Number: IRRB/16/22; Board Name: Comitato Etico IRCCS Sicilia.

Ancillary study of San Martino: Approval Number: 173/2021; Board Name: Comitato Etico Regionale della Liguria.

Ancillary study of Ca' Granda: Approval Number: 887_2020; Board Name: Comitato Etico Milano Area 2.

Ancillary study of Gemelli: Approval Number: 3614; Board Name: Comitato Etico della Fondazione Policlinico Universitario A. Gemelli IRCCS - Università Cattolica del Sacro Cuore.

Ancillary study of San Matteo: Approval Number: 2022-3.11/91 and 2022-3.11/493; Board Name: Comitato Etico Pavia.

Ancillary studiy of San Raffaele Roma: Approval Number: 21/21; Board Name: Comitato Etico IRCCS San Raffale Roma.

Update on Study Progress and Power Analysis: In its original design, the CV-PREVITAL study aimed to enrol approximately 80,000 subjects aged ≥45 years with no previous cardiovascular events. These participants were intended to be recruited from general practice clinics, pharmacies, or clinics of Scientific Institutes for Research, Hospitalization and Health Care (IRCCS). However, due to the challenges posed by the COVID-19 pandemic, which has fully engaged all parties involved in the study (primarily general practitioners, pharmacists, and IRCCS physicians), the planned activities of the study have been significantly delayed, especially in terms of participant enrollment. Despite these challenges, the study successfully recruited around 28,000 subjects, which is expected to be a sufficient number for evaluating the short-term primary endpoint. Specifically, to assess the short-term primary endpoint, a sample size of N=7895 per treatment arm is required, assuming a significance level of 0.05 and a power of 90%. Therefore, if the target of 16,000 subjects with completed follow-up is achieved, the study will have adequate power to reach the short-term primary endpoint. The estimation of the statistical power for the long-term endpoint will be carried out at the conclusion of the 7-year follow-up period when data regarding the actual dropout rate become available.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 45 years
* Have given their consent to participate in the study
* Subjects who have a smartphone

Exclusion Criteria:

* Current or previous cardiovascular disease (personal history of myocardial infarction, angina pectoris, arterial revascularization procedures, stroke, TIA, peripheral artery disease)
* Psychiatric disorders
* Participation in other clinical trials

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27520 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk as assessed by Modified Moli-Sani risk score in the Italian population | 12 months
  A score (modified Moli-Sani Risk Score) developed in the Italian population is used to analyze the efficacy of the intervention at 12 months. The risk score includes of blood pressure, HDL, LDL, triglyceride, blood glucose, overweight, physical activity, adhesion to Mediterranean diet and cigarette smoking. The modified Moli-Sani Risk Score may range from 0 to 100 and higher scores means higher risk. A 10% improvement in score between the baseline and final visit in the intervention group compared with the control group is assumed as indicator of intervention effectiveness.
Long-term CV clinical outcome at 7 years follow-up | 7 years
  Incidence of a composite outcome including myocardial infarction (MI), stroke, transient ischemic attack (TIA), peripheral artery disease or CV death. In case of multiple vascular events only the first is used in the analyses of composite outcome, whereas the specific outcome (e.g. MI or stroke) is used when the sub-analyses focused on cardio- or cerebrovascular events are run.

SECONDARY OUTCOMES:
Change of a combined endpoint including hypertension, diabetes, hypercholesterolemia | 12 months
  For each individual subject, the combined end-point will be calculated, at baseline and at month 12, as the number of variables out of target (according to last European Society of Cardiology guidelines), among blood pressure, HbA1c and blood cholesterol; therefore, its value will range between 0 and 3. The difference in the combined end-point between month 12 and baseline will be compared, between the two experimental groups, using Wilcoxon rank-sum test.
Systolic and diastolic blood pressure (mmHg) | 12 months
  Comparison of the mean change from baseline in blood pressure in the two experimental groups.
HDL-C, LDL-C, and triglycerides (mg/dL) | 12 months
  Comparison of the mean change from baseline in blood lipids in the two experimental groups.
HbA1c (%) | 12 months
  Comparison of the mean change from baseline in HbA1c in the two experimental groups.
Body weight (kg) | 12 months
  Comparison of the mean change from baseline in body weight in the two experimental groups.
Physical activity (IPAQ questionnaire) | 12 months
  Comparison of the mean change from baseline in levels of physical activity as assessed by the short version (9 items) of the IPAQ (International Physical Activity Questionnaire) in the two experimental groups.
Mediterranean diet adherence (PREDIMED questionnaire) | 12 months
  Comparison of the mean change from baseline in adherence to Mediterranean diet as assessed by PREDIMED (Prevention with Mediterranean Diet)" questionnaire in the two experimental groups. The PREDIMED score is a 14-item Mediterranean Diet adherence screener. Adherence is stratified in three categories: 1) low adherence (calculated score ≤5) 2) intermediate adherence (calculated score from 6 to 9), 3) high adherence (calculated score ≥10).
Mediterranean diet adherence (Moli-Sani questionnaire) | 12 months
  Comparison of the mean change from baseline in adherence to Mediterranean diet as assessed by the Moli-Sani study questionnaire in the two experimental groups. The Moli-Sani Mediterranean diet adherence score may range from 0 to 21, the latter reflecting the maximal adherence to Mediterranean diet.
Smoking status | 12 months
  Comparison of the mean change from baseline in cigarette smoking quantified by pack-years (number of packs of cigarettes smoked per day by the number of years the person has smoked) in the two experimental groups.
Alcohol intake | 12 months
  Comparison of the mean change from baseline in alcohol intake as assessed by PREDIMED (''Prevención con dieta mediterránea'') questionnaire in the two experimental groups.
Salt intake (MiniSal questionnaire) | 12 months
  Comparison of the mean change from baseline in salt intake as assessed by MiniSal questioner in the two experimental groups. The score may range from 0 to 11, the latter reflecting the maximal salt intake.
Stress (Perceived Stress Scale; PSS) | 12 months
  Comparison of the mean change from baseline in perceived stress as assessed by PSS (Perceived Stress Scale) in the two experimental groups. The PSS scale may range from 0 to 40 and higher values means higher perceived Stress.
Psychological distress (PHQ 4 questionnaire) | 12 months
  Comparison of the mean change from baseline in psychological distress as assessed by "Patient Health Questionnaire-4 (PHQ-4)" in the two experimental groups. The psychological distress PHQ-4 questionnaire may range from 0 to 12 and higher values means higher presence of the disorder.
Anxiety (PHQ 4 questionnaire) | 12 months
  Comparison of the mean change from baseline in anxiety as assessed by "Patient Health Questionnaire-4 (PHQ-4)" in the two experimental groups. The Anxiety PHQ-4 questionnaire may range from 0 to 6 and higher values means higher presence of the disorder.
Depression (PHQ 4 questionnaire) | 12 months
  Comparison of the mean change from baseline in depression as assessed by "Patient Health Questionnaire-4 (PHQ-4)" in the two experimental groups. The Depression PHQ-4 questionnaire may range from 0 to 6 and higher values means higher presence of the disorder.
Multidimensional Health Locus of Control Scale (MHLCS) - Internality | 12 months
  Comparison of the mean change from baseline in locus of control as assessed by "Multidimensional Health Locus of Control Scale (MHLCS)-Internality" in the two experimental groups. The MHLCS-Internality may range from 6 to 36 and higher values means greater subject's internal locus of control.
Multidimensional Health Locus of Control Scale (MHLCS) - Powerful Others Externality | 12 months
  Comparison of the mean change from baseline in locus of control as assessed by "Multidimensional Health Locus of Control Scale (MHLCS)-powerful-others-externality" in the two experimental groups. The MHLCS-powerful-others-externality may range from 6 to 36 and higher values means greater subject's external (dependent on others) locus of control.
Multidimensional Health Locus of Control Scale (MHLCS) - Chance Externality | 12 months
  Comparison of the mean change from baseline in locus of control as assessed by "Multidimensional Health Locus of Control Scale (MHLCS)-chance-externality" in the two experimental groups. The MHLCS-chance-externality may range from 6 to 36 and higher values means greater external (case-dependent) locus of control of the subject.
General Self Efficacy (GSE Scale) | 12 months
  Comparison of the mean change from baseline in general self-efficacy as assessed by "General Self Efficacy scale (GSE)" in the two experimental groups. The GSE scale may range from 10 to 40 and higher values mean greater self-efficacy perceived by the subject.
Risk propensity (RPS Scale) | 12 months
  Comparison of the mean change from baseline in risk propensity as assessed by "Risk Propensity Scale (RPS)" in the two experimental groups. The RPS scale may range from 7 to 63 and higher values mean greater propensity to take risks.
Sleep quality (Pittsburgh Sleep Quality Index) | 12 months
  Comparison of the mean change from baseline in sleep quality as assessed by "Pittsburgh Sleep Quality Index (PSQI)" in the two experimental groups. The PSQI may range from 0 to 21 and higher values mean lower sleep quality.
Subjects' adherence to data recording | 12 months
  The App developed in the project collects information to analyse the participant's compliance with the data recording activities suggested by the app itself (blood pressure and blood glucose measurements, etc.). The subjects' adherence to data recording activities suggested by the app is assessed as the proportion of activities actually accomplished over the activities suggested.
Interruptions in the use of the mHealth App | 12 months
  The App developed in the project provides functions able to assess the number of accesses over time of the participant and the actual use of the recommended tools. The interruptions in the use of the mHealth App is assessed as the number of weeks of lack of the actual use of the app.
Adherence to recommended therapies | 12 months
  As part of the project, information on current therapies are collected in the eCRF at both baseline and 12 months. This information, together with the clinical/anthropometric data collected on the same occasions, will make it possible to ascertain whether a possible discontinuation of one of the therapies recorded at baseline is due to a improvement in the participant's clinical profile or to poor compliance. A poor adherence to recommended therapies is assessed by computing the frequency of non-medically justified therapy discontinuation.
Cost/effectiveness of intervention | 7 years
  Incremental cost-effectiveness ratio (EUR/QALYs) calculated on the basis of costs related to intervention implementation (summation of costs of implementing and maintaining the IT platform, costs of the smartphone application, costs for healthcare professionals training for the use of the IT platform and costs for the involvement and education of participants) combined in an economic model with the QALYs (Quality Adjusted Life Years) modelled based on number of cardiovascular events (fatal and non-fatal) avoided during the seven years of follow-up.
House ownership as socioeconomic status indicator | 7 years
  House ownership as socio-economic factor relevant to cardiovascular risk - proportion of subjects who are homeowners.
Type of residence as socioeconomic status indicator | 7 years
  Type of residence as socio-economic factor relevant to cardiovascular risk - proportion of subjects living in urban (big or small city) or rural area.
Education as socioeconomic status indicator | 7 years
  Education as socio-economic factor relevant to cardiovascular risk - proportion of subjects with: (1) no education (2) elementary education (3) Lower middle school (4) Higher middle school (5) Graduate (6) postgraduate).
Employment status as socioeconomic status indicator | 7 years
  Employment status as socio-economic factor relevant to cardiovascular risk - proportion of subjects who: (1) have a full-time job, (2) work less than 5 days a week, (3) have a part-time job, (4) are disability pensioner, (5) are retired due to age limit, (6) are Partially retired, (7) are unemployed, (8) are Housewife.
Type of profession as socioeconomic status indicator | 7 years
  Type of profession as socio-economic factor relevant to cardiovascular risk - proportion of subjects who are: (1) professionals, (2) teachers, (3) large business owners, (4) small business owners, (5) services, (6) employees, (7) laborers, (8) farmers, (9) Other.
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) - history of hospitalization (questionnaire) | 7 years
  History of hospitalization for SARS-CoV-2 infection as a risk factor for vascular events - proportion of subjects hospitalized for SARS-CoV-2 infection among those who develop or not vascular events over the 7-year follow-up period.
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) - history of symptoms (questionnaire) | 7 years
  History of symptoms for SARS-CoV-2 infection as a risk factor for vascular events - proportion of subjects with symptoms for SARS-CoV-2 infection among those who develop or not vascular events over the 7-year follow-up period.
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) - history of asymptomatic disease (questionnaire) | 7 years
  History of asymptomatic SARS-CoV-2, documented by at least one positive swab, as a risk factor for vascular events - proportion of subjects with at least one positive swab for SARS-CoV-2 infection among those who do or do not develop vascular events during the 7-year follow-up period.
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) - history of vaccination (questionnaire) | 7 years
  History of vaccination against SARS-CoV-2 infection as a protective factor for vascular events - proportion of subjects with at least one dose of vaccination against SARS-CoV-2 infection among those who do or do not develop vascular events during the 7-year follow-up period.

OTHER OUTCOMES:
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): 12-month change in Oral Glucose Tolerance Test (OGTT) response in the CV-PREVITAL PREDIABETES sub-study cohort | 12 months
  Change compared to baseline in OGTT response in subjects of the CV-PREVITAL PREDIABETES sub-study cohort (1,000 subjects, including 200 with a diagnosis of type 2 diabetes mellitus (T2DM), 400 with a diagnosis of pre-diabetes and 400 normoglycaemic, randomized in the parent study).
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): 12-month change in insulinemia in the CV-PREVITAL PREDIABETES sub-study cohort | 12 months
  Change compared to baseline in insulinemia (µU/mL) in subjects of the CV-PREVITAL PREDIABETES sub-study cohort.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): 12-month change in high-sensitivity C-reactive protein (hs-CRP) in the CV-PREVITAL PREDIABETES sub-study cohort | 12 months
  Change compared to baseline in hs-CRP (mg/L) in subjects of the CV-PREVITAL PREDIABETES sub-study cohort.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): 12-month change in microalbuminuria in the CV-PREVITAL PREDIABETES sub-study cohort | 12 months
  Change compared to baseline in microalbuminuria [A/C ratio (mg/g creatinine)] in subjects of the CV-PREVITAL PREDIABETES sub-study cohort.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): 12-month change in Estimated Glomerular Filtration Rate (eGFR) in the CV-PREVITAL PREDIABETES sub-study cohort | 12 months
  Change compared to baseline in eGFR estimated by serum creatinine values (mg/dL) in subjects of the CV-PREVITAL PREDIABETES sub-study cohort.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): 12-month change in additional lipid parameters in the CV-PREVITAL PREDIABETES sub-study cohort | 12 months
  Change compared to baseline in fasting apolipoprotein B and lipoprotein(a) values (mg/dL) in subjects of the CV-PREVITAL PREDIABETES sub-study cohort.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): 12-month change in diabetes diagnosis in the CV-PREVITAL PREDIABETES sub-study cohort | 12 months
  Proportion of subjects who changed from a diagnosis of T2DM to a diagnosis of pre-diabetes or from a diagnosis of pre-diabetes to a diagnosis of normoglycemia, compared to the baseline examination.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): markers of carotid subclinical atherosclerosis in the CV-PREVITAL PREDIABETES sub-study cohort | month 0
  Comparison of baseline values of intima-media thickness (IMT) (mm); atherosclerotic plaque thickness (mm) and common carotid artery interadventitia diameter (mm) among normoglycemic, pre-diabetic and diabetic subjects.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): carotid plaque area in the CV-PREVITAL PREDIABETES sub-study cohort | month 0
  Comparison of baseline values of total plaque area (mm2) among normoglycemic, pre-diabetic and diabetic subjects.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): carotid plaque volume in the CV-PREVITAL PREDIABETES sub-study cohort | month 0
  Comparison of baseline values of total plaque volume (mm3) among normoglycemic, pre-diabetic and diabetic subjects.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): carotid wall echolucency in the CV-PREVITAL PREDIABETES sub-study cohort | month 0
  Comparison of baseline values of echolucency (grayscale levels, 0-255) of carotid biggest plaques and echolucency of carotid IMT among normoglycemic, pre-diabetic and diabetic subjects.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): endothelial function in the CV-PREVITAL PREDIABETES sub-study cohort | month 0
  Comparison of baseline values of endothelial function (reactive hyperemia index) measured by the EndoPAT device among normoglycemic, pre-diabetic and diabetic subjects.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): peripheral atherosclerosis in the CV-PREVITAL PREDIABETES sub-study cohort | month 0
  Comparison of the prevalence of an impaired Ankle Brachial Index (ABI) between normoglycemic, pre-diabetic and diabetic subjects.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): diabetic retinopathy in the CV-PREVITAL PREDIABETES sub-study cohort | month 0
  Comparison of the prevalence of diabetic retinopathy assessed by fundus retinography among normoglycemic, pre-diabetic and diabetic subjects.
Ancillary study of UO-1 (Centro Cardiologico Monzino IRCCS): Long-term clinical outcome in the CV-PREVITAL PREDIABETES sub-study cohort | 7 years
  Assessment of occurrence of cardiovascular events and overt diabetes over the 7-year follow-up period, depending on the length of time in prediabetes and the interaction of prediabetes with other risk factors (e.g. obesity, hypertension, hypertriglyceridemia, etc.).
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change of modifiable lifestyle-related cardiovascular risk factor such as smoking status, unhealthy diet and sedentary life in subjects of the Auxologico sub-study cohort | 12 months
  Difference between App and control group in the proportion of subjects with any of the following characteristics: low adherence to Mediterranean diet (PREDIMED/MEDAS ≤ 8), or with low physical activity according to IPAQ (International Physical Activity Questionnaire) [nov.2005] or to be current smoker at 1 year after randomization.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in 24-h blood pressure in hypertensive subjects | 12 months
  Comparison of the mean change from baseline in mean 24-h systolic BP in the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in body mass index in obese/overweight subjects | 12 months
  Comparison of the mean change from baseline in mean BMI (height (m) and weight (kg) combined (kg/m2)) of obese subjects of the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in sleep quality in subjects with sleep complaints | 12 months
  Comparison of the mean change from baseline in sleep quality as assessed by PSQI (Pittsburgh Sleep Quality Index) in the two experimental groups. The PSQI may range from 0 to 21 and higher values mean lower sleep quality.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in ambulatory blood pressure variables in hypertensive subjects | 12 months
  Comparison of the mean change from baseline in mean 24-h systolic blood pressure (SBP), 24-h diastolic blood pressure (DBP), day-time SBP, day-time DBP, night-time SBP, night-time DBP, SD 24-h SBP, SD 24-h DBP, SD day-time SBP, SD day-time DBP, SD night-time SBP, SD night-time DBP, in the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12- month change in dipping status in hypertensive subjects | 12 months
  Comparison of the mean change from baseline in the two experimental groups considering the dipping status defined as the difference between the mean systolic blood pressure in the day and mean systolic blood pressure during the night, expressed as a percentage of the day time mean, with the accepted normal between 10% and 20%.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in dietary salt intake in hypertensive subjects | 12 months
  Comparison of the mean change from baseline of 24h sodium urinary secretion in hypertensive subjects of the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change of cardiovascular risk (in hypertensive and obese/overweight subjects) | 12 months
  Comparison of the mean change from baseline in a cardiovascular risk score calculated according to clinical variables and biomarkers: Troponin I (cut off of 0.008 ng/mL), hs-CRP (cut off of 6.81 mg/L) and N terminal pro-BNP (cut off of 187 pg/mL) in the two experimental groups. The score will have a minimum of 0, high scores will mean high cardiovascular risk.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in microalbuminuria in hypertensive subjects | 12 months
  Comparison of the mean change from baseline in microalbuminuria [A/C ratio (mg/mmol)] in the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in creatinine in hypertensive subjects | 12 months
  Comparison of the mean change from baseline in creatinine (mg/dL) of the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in eGFR in hypertensive subjects | 12 months
  Comparison of the mean change from baseline in eGFR [estimated by serum creatinine values (mg/dL)] of the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in left ventricular hypertrophy in hypertensive subjects | 12 months
  Comparison of the mean change from baseline in presence/absence of left ventricular hypertrophy on ECG of the two experimental groups evaluated with Sokolow index and Cornell product.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month changes in acid uric level in hypertensive and obese/overweight subjects | 12 months
  Comparison of the mean change from baseline in acid uric level (mg/dL) of the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month changes in fasting insulinemia (in obese/overweight subjects) | 12 months
  Comparison of the mean change from baseline in fasting insulinemia (µU/mL) in the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month changes in fasting glucose levels (in obese/overweight subjects) | 12 months
  Comparison of the mean change from baseline in fasting glucose levels (mg/dL) in the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month changes in waist circumference (in obese/overweight subjects) | 12 months
  Comparison of the mean change from baseline in waist circumference (cm) in the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month changes in waist/hips ratio (in obese/overweight subjects) | 12 months
  Comparison of the mean change from baseline in waist/hips ratio in the two experimental groups.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in Epworth Sleepness scale (ESS) questionnaire score (in subjects with sleep complaints) | 12 months
  Comparison of the mean change from baseline in improvement in daytime sleepiness assessed by the Epworth Sleepness scale (ESS) questionnaire in the two experimental groups. The ESS has a minimum score of 4 and maximum of 24. Normal score ranges between 0 and 10.
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in obstructive sleep apnea (OSA) diagnosis (in subjects with sleep complaints) | 12 months
  Difference in the percentage of patients diagnosed with OSA at 1 year after randomization in the two experimental groups; diagnosis of OSA is usually defined by polysomnographic indices like the apnea-hypopnea index (AHI) where AHI <5/hour = normal; 5-14.9/hour = mild OSA; 15-29.9/hour = moderate OSA; and ≥30/hour = severe OSA
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in positive airway pressure (PAP) treatment (in subjects with OSA treated with PAP therapy) | 12 months
  Difference in the percentage of patients using positive airway pressure (PAP) devices at 1 year after randomization in the two experimental groups
Ancillary study of UO-2 (IRCCS Istituto Auxologico Italiano): 12-month change in PAP treatment usage (in subjects with OSA treated with PAP therapy) | 12 months
  Mean difference in the daily use of PAP devices at 1 year after randomization in the two experimental groups.
Ancillary study of UO-3 (Humanitas Research Hospital IRCCS): 12-month change from baseline of LDL-cholesterol levels (powered primary outcome) in the CV-PREVITAL coronary calcium score sub-study cohort | 12 months
  Comparison of 12-month change from baseline of LDL-cholesterol levels between subjects randomized to screening by CT scanning to determine the CAC (Coronary Artery Calcium) score or traditional risk factor assessment alone. CAC score is calculated by the Agatston method and by the determination of the volume of calcium. The Agatston method assesses the weighted sum of lesions with a density above 130 Hounsfield unit (HU), multiplying the area of calcium by a factor related to maximum plaque attenuation: factor 1=130-199 HU; factor 2= 200-299 HU; factor 3= 300-399 HU; and factor 4= ≥ 400 HU. The calcium volume is calculated by multiplying the number of voxels with calcification by the volume of each voxel, including all voxels with an attenuation > 130 HU. The study has 2x2 factorial design: subjects are first randomized 1:1 to app or usual care; each subject is then randomized 1:1 to CT scanning on top of traditional risk factor assessment or traditional risk factor assessment alone.
Ancillary study of UO-3 (Humanitas Research Hospital IRCCS): Rate of statin and aspirin therapy initiation in the CV-PREVITAL coronary calcium score sub-study cohort | 12 months
  Comparison of the rate of statin and aspirin therapy initiation between subjects randomized to screening by CT scanning or traditional risk factor assessment alone.
Ancillary study of UO-3 (Humanitas Research Hospital IRCCS):12-month change in lipid biomarkers in the CV-PREVITAL coronary calcium score sub-study cohort | 12 months
  Comparison of 12-month change in lipid biomarkers between subjects randomized to screening by CT scanning or traditional risk factor assessment alone.
Ancillary study of UO-3 (Humanitas Research Hospital IRCCS): SNPs associated with severe coronary artery calcification | 12 months
  Assessment of the predictive ability for severe coronary artery calcification of SNPs, either identified in previous genome wide association studies or newly identified in this study.
Ancillary study of UO-3 (Humanitas Research Hospital IRCCS): Incremental effectiveness, as assessed by healthy quality-adjusted life years (QALYs), of screening by CT scanning for coronary calcium score | 7 years
  Incremental effectiveness (QALYs) calculated by multiplying Years of Life x Utility Value, assuming a utility value (quality of life) between 1=perfect health and 0=death.
Ancillary study of UO-3 (Humanitas Research Hospital IRCCS): Incremental cost effectiveness ratio (ICERs) of screening by CT scanning for coronary calcium score | 7 years
  Incremental cost effectiveness ratios (ICERs) calculated by dividing incremental costs (EUR) by incremental effectiveness (QALYs).
Ancillary study of UO-3 (Humanitas Research Hospital IRCCS): long-term clinical outcome in the CV-PREVITAL coronary calcium score sub-study cohort | 7 years
  Comparison of 7-year major adverse cardiovascular and cerebrovascular events between subjects randomized to screening by CT scanning or traditional risk factor assessment alone.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in additional lipid parameters in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in apolipoprotein AI, apolipoprotein B and lipoprotein(a) values (mg/dL) in the sub-study cohort.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in glycemia in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in glycemia (mg/dL) in the sub-study cohort.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in Brain Natriuretic Peptide (BNP) in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in BNP (pg/mL) in the sub-cohort.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in creatinine evaluation in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in creatinine (mg/dL) of the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in eGFR evaluation in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in eGFR (mL/min/1.73 m2) of the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in microalbuminuria in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in microalbuminuria [A/C ratio (mg/g creatinine)] of the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in hs-CRP in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in hs-CRP (mg/dL) of the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in Interleukin 6 (IL-6) and Interleukin 1 beta (IL-1 beta) in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in IL-6 and IL-1 beta (pg/mL) of the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change in enzymatic tests in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in mean values (U/L) of the following enzymes: creatine phosphokinase (CPK), aspartate aminotransferase (AST), alanine transaminase (ALT) and gamma- glutamyltransferase (GGT) of the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change of Intimal-Media Thickness in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in the Intimal- Media Thickness (mm) measured by B-mode ultrasound of common in the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change of Intercellular adhesion molecule (ICAM) and Vascular Cell Adhesion Molecule (VCAM) in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in endothelial function measured by circulating levels of ICAM and VCAM (ng/mL) in the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change of Ankle Brachial Index in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in Ankle Brachial Index in the two experimental groups
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change of total 10 year cardiovascular risk in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in the cardiovascular risk measured by an algorithm named "SCORE" (Systematic COronary Risk Evaluation)) in the two experimental groups. The Score may range from 0 to 100 and higher scores means higher risk.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change of quality of life in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in the quality of life measured by the WHOQOL-Measuring Quality of Life questioner in the two experimental groups. The WHOQOL-Measuring Quality of Life questionnaire (World Health Organization Quality of Life - short version) is a questionnaire composed by 26 items that investigate four areas related to the quality of life (physical health, psychological, social relationships and environment). Answers are rated on a 5-point scale (from one to five, where one indicates disagree or never at all and five indicates completely agree or extremely; with the exception for items 3, 4, and 26 where the scoring need to be reverted). For each domain a mean score is obtained and then multiplied by 4 in order to transform the domain scores into a scaled score from 0 to 100. Overall, a higher score means a higher quality of life.
Ancillary study of UO-5 (IRCCS MultiMedica): 12-month change of psychological conditions risk in the sub-study cohort | 12 months
  Comparison of the mean change from baseline in psychological conditions measured through Mini Mental Status Test in the two experimental groups.
Ancillary study of UO-5 (IRCCS MultiMedica): Coronary Calcium Score (Hounsfield units) | 12 months
  Evaluation of Coronary Artery Calcium (CAC) score in patients with suspected familial hypercholesterolemia. CAC is detected by means of CT scanning as described by Agatston, who defined CAC as the product of the calcified plaque area and maximal calcium lesion density. Hecht et al., PMID=22672574 The CAC score is expressed with a number where 0 indicates the absence of coronary calcifications, from 1 to 400 the presence of coronary calcifications with a progressively higher risk (1-100 low, 101-400 moderate) and a score higher than 400 Hounsfield units a severe risk.
Ancillary study of UO-5 (IRCCS MultiMedica): Long-term clinical outcome in the sub-study cohort | 7 years
  Assessment of occurrence of cardiovascular events, diabetes and hypertension over the 7-year follow-up period.
Ancillary study of UO-6 (IRCCS Neuromed): 12-month change in hs-CRP in the CV-PREVITAL Neuromed sub-study cohort | 12 months
  Comparison of the mean change from baseline in hs-CRP (mg/L) in the CV-PREVITAL Neuromed sub-study cohort.
Ancillary study of UO-6 (IRCCS Neuromed): 12-month change in eGFR in the CV-PREVITAL Neuromed sub-study cohort | 12 months
  Comparison of the mean change from baseline in eGFR estimated by serum creatinine values (mg/dL) in the CV-PREVITAL Neuromed sub-study cohort.
Ancillary study of UO-6 (IRCCS Neuromed): 12-month change in additional dietary habits assessed in the CV-PREVITAL Neuromed sub-study cohort | 12 months
  Proportion of subjects who changed the consumption of ultraprocessed foods, according to the NOVA classification, compared to the baseline examination.
Ancillary study of UO-6 (IRCCS Neuromed): 12-month change in additional psycho-emotional indexes assessed in the CV-PREVITAL Neuromed sub-study cohort | 12 months
  Proportion of subjects who changed cognitive ability as measured by the Montreal cognitive assessment (MOCA) test, compared to the baseline.
Ancillary study of UO-6 (IRCCS Neuromed): Determinants of dietary changes in the CV-PREVITAL Neuromed sub-study cohort | 12 months
  Multivariable analyses of determinants associated with dietary changes over 12 months follow-up period.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline analysis of insulinemia in the CV-PREVITAL San Donato cohort | month 0
  Baseline analysis of insulinemia (µU/ml) in the CV PREVITAL sub-study cohort and specifically in individuals with comorbidities such as diabetes mellitus, overweight, obesity, abdominal obesity.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline analysis of Homocysteine in the CV-PREVITAL San Donato cohort | month 0
  Baseline analysis of homocysteine (µmol/L) in the CV PREVITAL sub-study cohort and specifically in individuals with comorbidities such as diabetes mellitus, overweight, obesity, abdominal obesity.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline analysis of CRP in the CV-PREVITAL San Donato cohort | month 0
  Baseline analysis of CRP (mg/dl) in the CV PREVITAL sub-study cohort and specifically in individuals with comorbidities such as diabetes mellitus, overweight, obesity, abdominal obesity.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline analysis of blood sodium and potassium levels in the CV-PREVITAL San Donato cohort | month 0
  Baseline analysis of blood levels of sodium (mmol/L) and potassium (mmol/L) in the CV PREVITAL sub-study cohort and specifically in individuals with comorbidities such as diabetes mellitus, overweight, obesity, abdominal obesity.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline analysis of sRAGE and IL-6 in the CV-PREVITAL San Donato cohort | month 0
  Baseline analysis of blood levels of soluble receptor for advanced glycation end products (sRAGE) (pg/ml) and interleukin-6 (IL-6) (pg/ml) in the CV PREVITAL sub-study cohort and specifically in individuals with comorbidities such as diabetes mellitus, overweight, obesity, abdominal obesity.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): 12-month change in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) in the CV-PREVITAL San Donato cohort | 12 months
  Changes compared to baseline of NT-proBNP (ng/L) in CV PREVITAL sub-study cohort including individuals with overweight, obesity, abdominal obesity.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): 12-month change in thyroid stimulating hormone (TSH) in the CV-PREVITAL San Donato cohort | 12 months
  Changes compared to baseline of TSH (µU/ml) in CV PREVITAL sub-study cohort including individuals with overweight, obesity, abdominal obesity.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline relative wall thickness (ratio), E/A (ratio), and E/e' (ratio) as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Baseline left ventricular relative wall thickness (ratio), i.e. the ratio of end-diastolic radius to wall thickness, as detected by transthoracic-echocardiogram; baseline E/A (ratio), i.e. the ratio of peak velocity blood flow from left ventricular relaxation in early diastole (the E wave) to peak velocity flow in late diastole caused by atrial contraction (the A wave), as detected by transthoracic-echocardiogram; baseline E/e' (ratio), i.e. the ratio of the peak early mitral inflow velocity (E) over the early diastolic mitral annular velocity (e'), as detected by transthoracic-echocardiogram.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline Heart Mass (g) in the CV-PREVITAL San Donato cohort as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Transthoracic-echocardiogram detected baseline mass (g).
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline end-diastolic volume (ml), end-systolic volume (ml) and left atrial volume (ml) as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Transthoracic-echocardiogram detected baseline end-diastolic volume (ml), end-systolic volume (ml) and left atrial volume (ml).
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline Ejection Fraction (EF; %) in the CV-PREVITAL San Donato cohort as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Transthoracic-echocardiogram detected baseline Ejection Fraction (EF; %).
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline maximal tricuspid regurgitation velocity (TRV max) (m/s) in the CV-PREVITAL San Donato cohort as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Transthoracic-echocardiogram detected baseline TRV max (m/s).
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline epicardial adipose tissue (mm) in the CV-PREVITAL San Donato cohort as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Transthoracic-echocardiogram detected baseline epicardial adipose tissue (mm), identified as the echo-free space between the outer wall of the myocardium and the visceral layer of pericardium).
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline Carotid Artery Ultrasound imagining markers (IMT and plaques thickness) as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Baseline carotid arteries intimal-media thickness (IMT, mm) and plaque thickness (mm) measured with carotid artery ultrasound.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline Carotid Artery Ultrasound imagining markers (Presence/absence of plaques) as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Presence/absence at baseline of carotid artery atherosclerotic plaques as detected by carotid artery ultrasound. An atherosclerotic lesion is considered plaque when its maximum thickness exceeds 1.5 mm.
Ancillary study of UO-7 (IRCCS Policlinico San Donato): Baseline Carotid Artery Ultrasound imagining markers (total plaque area) as predictor of cardiovascular events in the CV-PREVITAL San Donato cohort | 7 years
  Total baseline carotid plaque area (mm2). This variable is obtained by summing the areas of all atherosclerotic plaques visualized in the entire carotid tree by carotid ultrasound performed at baseline.
Ancillary study of UO-8 (Istituti Clinici Scientifici Maugeri IRCCS): Occurrence of cardiovascular events in the CV-PREVITAL MAUGERI sub-study cohort | 7 years
  Occurrence of cardiovascular events over the 7-year follow-up period depending on the length of time in physical activities programs.
Ancillary study of UO-8 (Istituti Clinici Scientifici Maugeri IRCCS): Occurrence of new diagnosis of organ damage in the CV-PREVITAL MAUGERI sub-study cohort | 7 years
  Occurrence new diagnosis of organ damage (silent ischemia) over the 7-year follow-up period depending on the length of time in physical activities programs.
Ancillary study of UO-8 (Istituti Clinici Scientifici Maugeri IRCCS): change in ankle brachial index (ABI) in the CV-PREVITAL MAUGERI sub-study cohort | 7 years
  Change in ABI over the 7-year follow-up period depending on the length of time in physical activities programs.
Ancillary study of UO-8 (Istituti Clinici Scientifici Maugeri IRCCS): change in coronary calcium score in the CV-PREVITAL MAUGERI sub-study cohort | 7 years
  Change in coronary calcium score as detected by CT scan over the 7-year follow-up period depending on the length of time in physical activities programs.
Ancillary study of UO-8 (Istituti Clinici Scientifici Maugeri IRCCS): change in markers of carotid damage in the CV-PREVITAL MAUGERI sub-study cohort | 7 years
  Change from baseline in carotid arteries intimal-media thickness (IMT, mm) and plaque thickness (mm) as detected by carotid artery ultrasound over the 7-year follow-up period depending on the length of time in physical activities programs and the interaction of physical activity with other risk factors (e.g. obesity, hypertension, hypertriglyceridemia, etc.).
Ancillary study of UO-9 (ISMETT): 12-month change in coronary calcium score in the two arms in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in CAC score (Coronary Artery Calcium score) as detected by CT scan in the two experimental groups. the CAC score is measured as described by Agatston, who defined CAC as the product of the calcified plaque area and maximal calcium lesion density. The lesion score is determined based on the maximal computed tomographic number in the following manner: 1= 130 to 199, 2= 200 to 299, 3 = 300 to 399, 4≥400 Hounsfield units. The latter means severe calcified plaque.
Ancillary study of UO-9 (ISMETT): 12-month change in myocardial fibrosis in the two arms in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in myocardial fibrosis as detected by cardiac magnetic resonance in the two experimental groups. Outcome measure is the Delayed Enhancement (DE) left ventricular (LV) mass expressed as percentage of total LV Mass, and obtained through a Late Gadolinium Enhancement cardiac magnetic resonance. A DE-LV Mass > 10% is considered abnormal.
Ancillary study of UO-9 (IRCCS ISMETT): 12-month change in biomarker of stress and heart failure in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in circulating levels (mg/dL) of creatinine, blood urea, nitrogen (BUN) and high sensitivity C-Reactive Protein (HS-CRP) (mg/dL) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): 12-month change in NT-proBN in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in NT-proBN (pg/mL) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): 12-month change in Na and K levels in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in levels of Na and K (mmol/L) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): 12-month change in homocysteine levels in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in levels of homocysteine (micromol/L) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): 12-month change in serum iron in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in serum iron (microg/dL) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): 12-month change in ferritin in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in levels of ferritin (ng/mL) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): 12-month change in transferrin in CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in levels of transferrin (g/L) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): platelet and white blood cell count in the CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in the absolute number (x10^3 per microliter) of white blood cell (WBC), platelets, neutrophils, lymphocytes, monocytes, eosinophils, and basophils in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): red blood cell (RBC) count in the CV-PREVITAL ISMETT cohort | 12 months
  Comparison of the mean change from baseline in the absolute number (x10^6 per microliter) of RBC in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): hemoglobin (Hb) in the CV-PREVITAL ISMETT sub-study cohort | 12 months
  Comparison of the mean change from baseline in values of Hb (g/dL) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): hematocrit (HCT) in the CV-PREVITAL ISMETT sub-study cohort | 12 months
  Comparison of the mean change from baseline in values of HCT (%) in the two experimental groups.
Ancillary study of UO-9 (IRCCS ISMETT): effect of specific cardiovascular risk factors on coronary calcium score in the CV PREVITAL ISMETT cohort | 12 months
  Between group (usual-care and intervention) comparison of 12-months change in CAC score (Coronary Artery Calcium score) after stratification of the cohort according to specific cardiovascular risk factors (e.g. obesity, hypertension, diabetes etc). the CAC score is measured as described by Agatston, who defined CAC as the product of the calcified plaque area and maximal calcium lesion density. The lesion score is determined based on the maximal computed tomographic number in the following manner: 1= 130 to 199, 2= 200 to 299, 3 = 300 to 399, 4≥400 Hounsfield units. The latter means severe calcified plaque.
Ancillary study of UO-9 (IRCCS ISMETT): effect of specific cardiovascular risk factors on myocardial fibrosis in the CV PREVITAL ISMETT cohort | 12 months
  Between group (usual-care and intervention) comparison of 12-months change in myocardial fibrosis as detected by cardiac magnetic resonance after stratification of the cohort according to specific cardiovascular risk factors (e.g. obesity, hypertension, diabetes etc).
Ancillary study of UO-9 (IRCCS ISMETT): effect of specific cardiovascular risk factors on biomarkers of stress and heart failure in the CV PREVITAL ISMETT cohort | 12 months
  Between group (usual-care and intervention) comparison of 12-months change in circulating levels (mg/dL) of creatinine, blood urea and CRP (mg/dL) after stratification of the cohort according to specific cardiovascular risk factors (e.g. obesity, hypertension, diabetes etc).
Ancillary study of UO-10 (Ospedale Policlinico San Martino IRCCS): Prevalence of abdominal aortic aneurysms in the CV-PREVITAL San Martino sub-study cohort | month 0
  Measurement of maximum diameter (mm) of abdominal aorta arteries by ultrasound in 1500 male subjects aged ≥ 45 years enrolled for primary prevention to identify eventual presence of aneurysms and estimate prevalence.
Ancillary study of UO-10 (Ospedale Policlinico San Martino IRCCS): Prevalence of iliac artery aneurysms in the CV-PREVITAL San Martino sub-study cohort | month 0
  Measurement of maximum diameter (mm) of iliac arteries by ultrasound in 1500 male subjects aged ≥ 45 years enrolled for primary prevention to identify eventual presence of aneurysms and estimate prevalence.
Ancillary study of UO-10 (Ospedale Policlinico San Martino IRCCS): Prevalence of carotid artery stenosis in the CV-PREVITAL San Martino sub-study cohort. | month 0
  Assessment of the prevalence of carotid artery stenosis in 500 male subjects aged ≥ 45 years enrolled for primary prevention.
Ancillary study of UO-10 (Ospedale Policlinico San Martino IRCCS): risk stratification for cardiovascular disease in the CV-PREVITAL San Martino sub-study cohort. | month 0
  Measurement of the intima-media thickness of the supra-aortic trunks to increase the early identification of individuals prone to develop atherosclerosis and risk stratification for cardiovascular disease.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in markers of carotid damage (intimal-media thickness and plaques thickness) in the two arms in CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in carotid arteries intimal-media thickness (IMT, mm) and plaque thickness (mm) as detected by carotid artery ultrasound in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in markers of carotid damage (Presence/absence of plaques) in the two arms in CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in the prevalence of carotid artery atherosclerotic plaques as detected by carotid artery ultrasound in the two experimental groups. An atherosclerotic lesion is considered plaque when its maximum thickness exceeds 1.5 mm.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in Fibroscan CAP Score as a non-invasive biomarker of liver damage in the CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in the amount of hepatic fat estimated non-invasively by using Fibroscan (CAP Score, dB/m) in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in Fibrosis-4 Index (FIB-4) as non-invasive biomarker of liver damage in the CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in the hepatic fibrosis stage (FIB-4 Index) estimated non-invasively by using Fibroscan (Liver Stiffness Measurement - LSM, kPa) in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in circulating biomarker of lipotoxicity (Interleukin-32) in the CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in interleukin-32 (IL-32, pg/mL) blood levels, as a biomarker of lipotoxicity in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in microalbuminuria in the CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in microalbuminuria urine's levels as a biomarker of renal injury (mg/L) in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in enzymatic tests in the CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in mean values (U/L) of aspartate aminotransferase (AST), alanine transaminase (ALT) and gamma-glutamyltransferase in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): 12-month change in insulinemia in the CV-PREVITAL blood donor sub-study cohort | 12 months
  Comparison of the mean change from baseline in Insulinemia blood levels as biomarker of insulin resistance (microU/mL) in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): characterization of the coagulation balance in the CV-PREVITAL blood donor sub-study cohort | month 0
  Comparison of the baseline levels (%) of von Willebrand Factor Antigen, Protein C and Factor VIII in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): D-Dimer levels in the CV-PREVITAL blood donor sub-study cohort | month 0
  Comparison of baseline D-Dimer levels (ng/ml) in the two experimental groups.
Ancillary study of UO-11 (IRCCS Ca' Granda): 7-year change in taxonomic characterization of the intestinal microbiome in feces in a subsample of 200 participants | 7 years
  Characterization of the intestinal microbiome in feces in a subsample of 200 participants by conducting a taxonomic analysis, with particular attention to Bacteroidetes/Firmicutes ratio.
Ancillary study of UO-11 (IRCCS Ca' Granda): 7-year change in characterization of the intestinal microbiome in feces in a subsample of 200 participants | 7 years
  Characterization of the microbiome metagenomic functional profile in a subsample of 200 participants.
Ancillary study of UO-11 (IRCCS Ca' Granda): 7-year change in the intestinal microbiome in feces in a subsample of 200 participants (TMAO) | 7 years
  Characterization of the intestinal microbiome in feces in a subsample of 200 participants by evaluation of TMAO serum levels.
Ancillary study of UO-11 (IRCCS Ca' Granda): 7-year change in characterization of the intestinal microbiome in feces in a subsample of 200 participants (branched-chain amino acid, BCAAs) | 7 years
  Characterization of the intestinal microbiome in feces in a subsample of 200 participants by evaluation of branched-chain amino acid (BCAAs).
Ancillary study of UO-11 (IRCCS Ca' Granda): 7-year change in characterization of the intestinal microbiome in feces in a subsample of 200 participants (aromatic amino acid, AAAs) | 7 years
  Characterization of the intestinal microbiome in feces in a subsample of 200 participants by evaluation of aromatic amino acid (AAAs).
Ancillary study of UO-12 (IRCCS Gemelli): 12-month change in thickness of the medium-intimal complex of the common carotid in the CV-PREVITAL Inflammation and Microbiota sub-study cohort | 12 months
  Comparison of the mean change from baseline in carotid imaging (Intimal- Media Thickness measured in plaque-free areas of common carotid arteries) in the two experimental groups.
Ancillary study of UO-12 (IRCCS Gemelli): 12-month change in additional lipid parameters in the CV-PREVITAL-Inflammation and Microbiota sub-study cohort | 12 months
  Comparison of the mean change from baseline in lipoprotein(a) and oxLDL values (ng/dL) in the two experimental groups.
Ancillary study of UO-12 (IRCCS Gemelli): 12-month change in hs-CRP in the CV-PREVITAL Inflammation and Microbiota sub-study cohort | 12 months
  Comparison of the mean change from baseline in hs-CRP (mg/L) in the two experimental groups.
Ancillary study of UO-12 (IRCCS Gemelli): 12-month change in inflammatory mediators in the CV-PREVITAL-Inflammation and Microbiota sub-study cohort | 12 months
  Comparison of the mean change from baseline in plasma IL1beta, IL-18, IL-6, IL-10, TNF-alpha, and LPS values (pg/mL) in the two experimental groups.
Ancillary study of UO-12 (IRCCS Gemelli): 12-month change in serum levels of trimethylamine oxide (TMAO) in the CV-PREVITAL Inflammation and Microbiota sub-study cohort | 12 months
  Comparison of the mean change from baseline serum levels of TMAO (micromol/L) in the two experimental groups.
Ancillary study of UO-12 (IRCCS Gemelli): 12-month change in intestinal microbiome composition and intestinal permeability in the CV-PREVITALInflammation and Microbiota sub-study cohort | 12 months
  Change compared to baseline data of intestinal microbiome composition with Next Generation Sequencing (NGS) technology to identify alteration in the composition of the intestinal microbiome, both at a taxonomic and bacterial functional level. Change compared to baseline of zonulin serum level, a marker of intestinal permeability.
Ancillary study of UO-12 (IRCCS Gemelli):Long-term clinical outcome in the CV-PREVITAL Inflammation and Microbiota sub-study cohort | 7 years
  Assessment of occurrence of cardiovascular events over the 7-year follow-up period, depending on the significant biomarkers variation and microbiome composition detected in the CV-PREVITAL Inflammation and Microbiota sub-study (OxLDL, TMAO, Zonulin, bacterial intestinal composition, etc.).
Ancillary study of UO-13 (IRCCS San Matteo): NGS multigene analysis for the early diagnosis of diabetes | 7 years
  Prevalence of likely pathogenic and pathogenic variants classified according to ACMG criteria in genes related with diabetes in non-diabetic, pre-diabetic and diabetic subjects is analyzed by NGS panels of genes linked to monogenic diabetes in subjects of the San Matteo cohort and in subjects recruited by the IRCCS Monzino within the CV-PREVITAL PREDIABETES sub-study. DNA is collected from white blood cells. The gene prevalence is calculated as the ratio between patients carrying pathogenic variants and all patients of the studied cohort.
Ancillary study of UO-13 (IRCCS San Matteo): NGS multigene analysis for the diagnosis of familial dyslipidemia | 7 years
  Prevalence of likely pathogenic and pathogenic variants classified according to ACMG criteria in genes related with familial hypercholesterolemia in subjects with diagnosis of hypercholesterolemia is analyzed by NGS panels of genes associated with familial hypercholesterolemia. The studied subjects are from the San Matteo cohort and from patients recruited by the IRCCS Monzino within the CV-PREVITAL PREDIABETES sub-study. DNA is collected from white blood cells.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of physical activity in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in levels of physical activity as assessed by IPAQ (International Physical Activity Questionnaire) in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): amount of daily physical activity in the CV-PREVITAL Exercise sub-study cohort | 3 months and 6 months
  Change from baseline in the amount of daily physical activity measured through an accelerometer app in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of Mediterranean diet adherence by MDS questioner in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in adherence to Mediterranean diet as assessed by MDS (Mediterranean diet Scale)" questioner in the two experimental groups. The MDS scale may range from 0 to 55 and higher scores means higher Mediterranean diet adherence.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of Mediterranean diet adherence by PREDIMED questioner in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in adherence to Mediterranean diet as assessed by PREDIMED (''Prevención con dieta mediterránea'') questioner in the two experimental groups. The PREDIMED score may range from 0 to 14 and higher scores means higher Mediterranean diet adherence.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of Mediterranean diet adherence by Moli-Sani questioner in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in adherence to Mediterranean diet as assessed by the Moli-Sani study questioner in the two experimental groups. The Moli-Sani score may range from 0 to 21 and higher scores means higher Mediterranean diet adherence.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): salt intake in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in salt intake as assessed by MiniSal questionnaire in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of alcohol intake in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in alcohol intake as assessed by PREDIMED (''Prevención con dieta mediterránea'') questioner in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of stress (Perceived Stress Scale; PSS) in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in perceived stress as assessed by Perceived Stress Scale (PSS) in the two experimental groups. The PSS scale may range from 0 to 40 and higher values means higher perceived Stress.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of psychological distress (PHQ 4 questioner) in the CV-PREVITAL Exercise sub- study cohort | 6 months
  Comparison of the mean change from baseline in psychological distress as assessed by "Patient Health Questioner-4 (PHQ-4)" in the two experimental groups. The psychological distress PHQ-4 questioner may range from 0 to 12 and higher values means higher presence of the disorder.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of anxiety (PHQ 4 questioner) in the CV-PREVITAL Exercise sub- study cohort | 6 months
  Comparison of the mean change from baseline in anxiety as assessed by "Patient Health Questioner-4 (PHQ-4)" in the two experimental groups. The Anxiety PHQ-4 questioner may range from 0 to 6 and higher values means higher presence of the disorder.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of depression (PHQ 4 questioner) in the CV-PREVITAL Exercise sub- study cohort | 6 months
  Comparison of the mean change from baseline in depression as assessed by "Patient Health Questioner-4 (PHQ-4)" in the two experimental groups. The Depression PHQ-4 questioner may range from 0 to 6 and higher values means higher presence of the disorder.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of General Self Efficacy (GSE Scale) in the CV-PREVITAL Exercise sub- study cohort | 6 months
  Comparison of the mean change from baseline in general self-efficacy as assessed by "General Self Efficacy scale (GSE)" in the two experimental groups. The GSE scale may range from 10 to 40 and higher values mean greater self-efficacy perceived by the subject.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of Multidimensional Health Locus of Control Scale (MHLCS) - Internality in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in locus of control as assessed by "Multidimensional Health Locus of Control Scale (MHLCS)-Internality" in the two experimental groups. The MHLCS-Internality may range from 6 to 36 and higher values means greater subject's internal locus of control.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of Multidimensional Health Locus of Control Scale (MHLCS) - Powerful Others Externality in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in locus of control as assessed by "Multidimensional Health Locus of Control Scale (MHLCS)-powerful-others-externality" in the two experimental groups. The MHLCS-powerful-others-externality may range from 6 to 36 and higher values means greater subject's external (dependent on others) locus of control.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of Multidimensional Health Locus of Control Scale (MHLCS) - Chance Externality in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in locus of control as assessed by "Multidimensional Health Locus of Control Scale (MHLCS)-chance-externality" in the two experimental groups. The MHLCS-chance-externality may range from 6 to 36 and higher values means greater external (case-dependent) locus of control of the subject.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of Risk propensity in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in risk propensity as assessed by "Risk Propensity Scale (RPS)" in the two experimental groups. The RPS scale may range from 7 to 63 and higher values mean greater propensity to take risks.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of sleep quality in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in sleep quality as assessed by "Pittsburgh Sleep Quality Index (PSQI)" in the two experimental groups. The PSQI may range from 0 to 21 and higher values mean lower sleep quality.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of HDL-C, LDL-C, triglycerides and blood glucose in the CV- PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in fasting blood lipids and glucose levels (mg/dl) in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): 6 month-evaluation of HbA1c in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in HbA1c (%) in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): red blood cell (RBC) count in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in the absolute number (x10^6 per microliter) of RBC in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): platelet and white blood cell count in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in the absolute number (x10^3 per microliter) of white blood cell (WBC), platelets, neutrophils, lymphocytes, monocytes, eosinophils, and basophils in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): differential WBC count in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in the percent (%) of neutrophils, lymphocytes, monocytes, eosinophils, and basophils in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): hematocrit (HCT) and RBC Distribution Width (RDW) in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in values of HCT and RDW (%) in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): mean corpuscular volume (MCV) and mean platelet volume (MPV) in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in values of MCV and MPV (fL) in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): hemoglobin (Hb) and mean corpuscular hemoglobin concentration (MCHC) in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in values of Hb and MCHC (g/dL) in the two experimental groups.
Ancillary study of UO-14 (IRCCS San Raffaele Roma): mean corpuscular hemoglobin (MCH) in the CV-PREVITAL Exercise sub-study cohort | 6 months
  Comparison of the mean change from baseline in values of MCH (pg) in the two experimental groups.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Pompilio, Professor, Principal Investigator — Centro Cardiologico Monzino IRCCS; Gianfranco Parati, Professor, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (32):
- Italy (32):
  - Nucleo Cure Primarie Val Pescara, Scafa, Abruzzo
  - Progetto Salute Soc. Coop, Martano, Apulia
  - Panacea Medical Group, Reggio Calabria, Calabria
  - Samnium Medica, Benevento, Campania
  - MEDINCO', Salerno, Campania
  - Magna Grecia, Salerno, Campania
  - Meditem, Carpi, Emilia-Romagna
  - MAF, Pradamano, Friuli Venezia Giulia
  - IRCCS Neuromed, Pozzilli, Isernia
  - Arvamed, Rome, Lazio
  - IRCCS San Raffaele Roma, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - MediCoop Genova, Genoa, Liguria
  - Ospedale Policlinico San Martino IRCCS, Genoa, Liguria
  - Medici Insubria, Appiano Gentile, Lombardy
  - IML, Bergamo, Lombardy
  - GST, Legnano, Lombardy
  - CMMC, Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Centro Cardiologico Monzino, Milan, Lombardy
  - Istituto Auxologico Italiano IRCCS, Milan, Lombardy
  - Cosma 2000, Mozzate, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Lombardy
  - Humanitas Research Hospital IRCCS, Rozzano, Lombardy
  - IRCCS Policlinico San Donato, San Donato Milanese, Lombardy
  - IRCCS MultiMedica SpA, Sesto San Giovanni, Lombardy
  - CMMG Soresina, Soresina, Lombardy
  - IRCCS Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione (ISMETT), Palermo, Sicily
  - ARS Medica, Seravezza, Tuscany
  - Medici 2000, Siena, Tuscany
  - Medigen Salute, Padua, Veneto

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing plan is under definition

REFERENCES:
- [Derived] Baldassarre D, Iacoviello L, Baetta R, Roncaglioni MC, Condorelli G, Remuzzi G, Gensini G, Frati L, Ricciardi W, Conaldi PG, Uccelli A, Blandini F, Bosari S, Scambia G, Fini M, Di Malta A, Amato M, Veglia F, Bonomi A, Klersy C, Colazzo F, Pengo M, Gorini F, Auteri L, Ferrante G, Baviera M, Ambrosio G, Catapano A, Gialluisi A, Malavazos AE, Castelvecchio S, Corsi-Romanelli MM, Cardani R, La Rovere MT, Agnese V, Pane B, Prati D, Spinardi L, Liuzzo G, Arbustini E, Volterrani M, Visconti M, Werba JP, Genovese S, Bilo G, Invitti C, Di Blasio A, Lombardi C, Faini A, Rosa D, Ojeda-Fernandez L, Foresta A, De Curtis A, Di Castelnuovo A, Scalvini S, Pierobon A, Gorini A, Valenti L, Luzi L, Racca A, Bandi M, Tremoli E, Menicanti L, Parati G, Pompilio G; CV-PREVITAL Study Group. Rationale and design of the CV-PREVITAL study: an Italian multiple cohort randomised controlled trial investigating innovative digital strategies in primary cardiovascular prevention. BMJ Open. 2023 Jul 14;13(7):e072040. doi: 10.1136/bmjopen-2023-072040. PMID 37451717